CLINICAL TRIAL: NCT06843382
Title: Real-World Comparative Effects of Teriflunomide and Dimethyl Fumarate on Physical and Cognitive Fatigability in Multiple Sclerosis: The ROOF-MS Multicenter Prospective Cohort Study
Brief Title: Real-world Experience of Oral Agents On Fatigability in Multiple Sclerosis
Acronym: ROOF-MS
Status: Not yet recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Collaborators: Sakarya University (Other); Kocaeli University (Other); Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Fatih Yetkin, Principal Investigator, Head of Multiple Sclerosis Unit of Erciyes University, TC Erciyes University
Other Study IDs: ROOF-MS
Record Dates: First submitted 2025-01-22; First posted 2025-02-25 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Teriflunomide; Fatigability; Real-world study
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Teriflunomide Cohort: Participants with relapsing multiple sclerosis who initiate teriflunomide as part of routine clinical care. Individuals in this cohort undergo standardized assessments of physical and cognitive fatigability, functional performance, clinical status, patient-reported outcomes, and routinely obtained MRI findings at baseline and at 3, 6, 9, and 12 months. No experimental treatment is administered, and all therapeutic decisions remain under the responsibility of the treating physician.
- Dimethyl Fumarate Cohort: Participants with relapsing multiple sclerosis who initiate dimethyl fumarate as part of routine clinical care. Individuals in this cohort complete standardized evaluations of physical and cognitive fatigability, functional performance, clinical status, patient-reported outcomes, and routinely acquired MRI measures at baseline and at 3, 6, 9, and 12 months. No experimental intervention is provided, and all treatment decisions are made independently by the treating physician.

SUMMARY:
This multicenter, prospective, real-world study evaluates how two commonly used oral disease-modifying therapies-teriflunomide and dimethyl fumarate-affect physical and cognitive fatigability in adults with multiple sclerosis (MS). Fatigability refers to an objective decline in physical or cognitive performance during sustained activity and represents a major barrier to daily functioning for many individuals with MS.

Participants starting either teriflunomide or dimethyl fumarate as part of routine clinical care will be followed for 12 months at regular visits (baseline, 3, 6, 9, and 12 months). At each visit, standardized assessments will measure walking endurance, gait performance, hand function, and information-processing speed. Patient-reported outcomes about fatigue, mood, quality of life, and daily functioning will also be collected. Brain MRI scans performed as part of usual care will be reviewed to document disease activity.

The goal of the ROOF-MS study is to understand whether these two therapies differ in their impact on physical and cognitive fatigability, functional outcomes, symptom burden, and real-world treatment adherence. Because this is an observational study, no experimental treatments are given, and all clinical decisions remain the responsibility of the treating physicians.

By examining fatigability in everyday clinical settings, this study aims to generate evidence that can help patients, families, and health care providers make more informed treatment decisions.

DETAILED DESCRIPTION:
This investigator-initiated, multicenter, prospective observational cohort study examines longitudinal changes in physical and cognitive fatigability among adults with multiple sclerosis (MS) initiating teriflunomide or dimethyl fumarate as part of routine clinical care. The study integrates standardized fatigability assessments into real-world clinical workflows across participating neurology centers.

Fatigability represents an objective performance decline during sustained motor or cognitive activity and provides information that is complementary to subjective fatigue ratings. To quantify physical fatigability, the study applies a structured 6-Minute Walk Test protocol in which distance covered during each minute is recorded. The primary physical fatigability index (DWI6-1) is calculated as the percentage change between the first and sixth minutes, enabling sensitive detection of time-dependent gait deterioration. Cognitive fatigability is quantified via a timed Symbol Digit Modalities Test procedure in which correct responses are recorded at three consecutive 30-second intervals. The Cognitive Fatigability Index (CFI-SDMT) reflects the proportional change between early and late test performance. Both indices allow continuous modeling of longitudinal trajectories and group differences.

All assessments are performed at baseline (within 30 days of treatment initiation) and at months 3, 6, 9, and 12. Functional performance measures (6MWT total distance, Timed 25-Foot Walk, Nine-Hole Peg Test), clinical evaluations (EDSS), patient-reported outcomes (FIS, TSQM, HADS), and MRI findings obtained during routine care are incorporated to contextualize patterns of fatigability. Test administration is standardized across centers through written manuals and joint training sessions. To minimize diurnal variability, fatigability tests are scheduled at approximately the same time of day for each participant.

Because the study is non-interventional, treatment decisions-including drug choice, dosing, and management of side effects-are determined solely by treating physicians. Data are recorded in a secure electronic capture platform using coded identifiers, with center-level access restrictions and prospective time-locked entry to maintain data integrity. All analyses follow a predefined statistical plan using mixed-effects modeling with participant- and center-level random effects to account for repeated measures and between-center heterogeneity.

This study aims to clarify real-world differences in fatigability trajectories between teriflunomide and dimethyl fumarate and to determine how these trajectories relate to functional performance, symptomatic burden, radiological disease activity, and treatment adherence in routine MS care.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing Multiple Sclerosis (RRMS or active SPMS) diagnosis, confirmed according to the 2017 revised McDonald criteria.
* 18 years or older at the time of enrollment.
* Newly initiated teriflunomide treatment as part of routine clinical care.
* Ambulatory status (EDSS ≤ 7.0), capable of completing study assessments.
* Ability and willingness to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Diagnosis of Primary Progressive Multiple Sclerosis (PPMS).
* Severe comorbidities affecting mobility or cognitive function (e.g., advanced cardiovascular, pulmonary, or neuromuscular disease).
* Neurological or psychiatric conditions that prevent cognitive testing (e.g., advanced cognitive impairment, untreated severe depression).
* Severe upper extremity motor dysfunction, limiting 9-Hole Peg Test (9-HPT) or Symbol Digit Modalities Test (SDMT) completion.
* Pregnancy or breastfeeding at the time of enrollment.
* Inability to comply with study visits at baseline, 3 months, 6 months, and 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 18 years or older with a confirmed diagnosis of relapsing Multiple Sclerosis (MS), including relapsing-remitting MS (RRMS) and active secondary progressive MS (SPMS), according to the 2017 revised McDonald criteria. Participants will be selected from routine clinical settings where teriflunomide has been prescribed as part of standard care. Eligible individuals must be ambulatory, with an Expanded Disability Status Scale (EDSS) score of 7.0 or lower, and capable of performing the 6-Minute Walk Test (6MWT). This population will represent a real-world cohort reflective of patients receiving teriflunomide in typical clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Walking Fatigability Index | Assessments will be conducted at baseline, at three months, at six months, and at twelve months following treatment initiation.
  Walking fatigability will be quantified using the Distance Walk Index (DWI), calculated with the following formula:
  DWI=(Distance at minute 6-Distance at minute 1Distance at minute 1)×100 DWI=(Distance at minute 1Distance at minute 6-Distance at minute 1 )×100
  A DWI decline of >10% will be classified as abnormal, based on prior relapsing-remitting MS studies.
  Unit of Measurement: Percentage (%) Time Frame: Baseline, 3 months, 6 months, and 12 months Higher Values Indicate: Better walking endurance (lower fatigability)
Cognitive Fatigability Index | Baseline, 3 months, 6 months, and 12 months
  Cognitive fatigability will be quantified using the Cognitive Fatigability Index (CFI), calculated with the following formula:
  CFI=(SDMT3-SDMT1SDMT1)×100 CFI=(SDMT1SDMT3-SDMT1 )×100
  A negative CFI value will indicate cognitive fatigability, with a decline greater than 10% classified as abnormal.
  Unit of Measurement: Percentage (%) Higher Values Indicate: Better cognitive endurance (lower fatigability)

SECONDARY OUTCOMES:
Walking Performance | Baseline, 3 months, 6 months, and 12 months
  Walking performance will be assessed using the 6-Minute Walk Test (6MWT). The total distance walked (meters) and walking speed (meters per minute, m/min) will be recorded.
  Unit of Measurement: Meters (m), Meters per minute (m/min) Higher Values Indicate: Better walking endurance
Radiological Outcomes | Radiological outcomes will be assessed at three time points: baseline (prior to treatment initiation), 6 months after starting treatment, and 12 months after starting treatment.
  Radiological outcomes will assess MRI changes at baseline, 6 months, and 12 months to evaluate disease progression and lesion activity in MS.
  T2 Lesions: Total number of T2-weighted hyperintense lesions. Gadolinium-Enhancing Lesions: Presence and count of Gd-enhancing lesions. New Lesions: Number of newly developed brain and spinal cord lesions. Upper Cervical Spinal Lesions: Presence of lesions in C1-C4 spinal cord region. Brainstem Lesions: Identification of lesions in the brainstem.
  Unit: Lesion count per MRI scan Higher Values Indicate: Increased disease activity
Walking Endurance | Baseline, 3 months, 6 months, and 12 months
  Walking endurance will be assessed using the 6-Minute Walk Test (6MWT). Participants will walk at their fastest pace to cover the maximum distance within six minutes, following the standardized protocol by Goldman et al. The total distance walked (meters) will be recorded as the primary measure of endurance.
  Unit of Measurement: Meters (m) Higher Values Indicate: Better walking endurance (lower fatigability)
Processing Speed and Attention | Baseline, 3 months, 6 months, and 12 months
  Processing speed and sustained attention will be assessed using the Symbol Digit Modalities Test (SDMT), a validated neurocognitive test. Participants will complete the SDMT in a 90-second timed format following the standardized protocol.
  Correct responses will be recorded at three consecutive 30-second intervals, and the total number of correct responses will be reported.
  Unit of Measurement: Number of correct responses Higher Values Indicate: Better cognitive processing speed and sustained attention
Hand Coordination and Dexterity | Baseline, 3 months, 6 months, and 12 months
  Hand coordination and dexterity will be evaluated using the 9-Hole Peg Test (9-HPT) for both hands. The time (in seconds) required to complete the task will be recorded.
  Unit of Measurement: Seconds (s) Higher Values Indicate: Worse dexterity
Fatigue Severity | Baseline, 3 months, 6 months, and 12 months
  Fatigue severity will be evaluated using the Fatigue Impact Scale (FIS), a validated patient-reported measure assessing the perceived impact of fatigue on cognitive, physical, and psychosocial functioning. Participants rate the extent to which fatigue has affected daily activities during the previous month. Higher scores indicate greater fatigue-related impact.
  Time Frame: Baseline, Month 3, Month 6, Month 9, Month 12 Type of Outcome: Patient-Reported Outcome Measure Method of Aggregation: Mean change from baseline and longitudinal trajectory over 12 months.
Treatment Satisfaction | Baseline, 3 months, 6 months, and 12 months
  Treatment satisfaction will be measured using the Treatment Satisfaction Questionnaire for Medication (TSQM). This instrument assesses satisfaction with medication across different domains (effectiveness, side effects, convenience, and global satisfaction).
  Unit of Measurement: TSQM Score (range to be specified) Higher Values Indicate: Greater treatment satisfaction
Anxiety and Depression | Baseline, 3 months, 6 months, and 12 months
  Anxiety and depression symptoms will be assessed using the Hospital Anxiety and Depression Scale (HADS), which consists of two subscales:
  HADS-Anxiety (HADS-A): Scores range from 0 to 21, with higher scores indicating greater anxiety.
  HADS-Depression (HADS-D): Scores range from 0 to 21, with higher scores indicating greater depressive symptoms.
  Unit of Measurement: HADS Score (0-21 per subscale) Higher Values Indicate: Greater anxiety or depression

OTHER OUTCOMES:
Safety outcomes | From enrollment through study completion at 12 months, with assessments at baseline, 3 months, 6 months, and 12 months
  The safety profile of teriflunomide will be assessed by monitoring the incidence, severity, and type of adverse events (AEs), including laboratory abnormalities, hair thinning or loss, and other treatment-related side effects. Serious adverse events (SAEs) will be categorized according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0), assessing their severity and relationship to treatment.
  Unit: Incidence count of AEs/SAEs
  Higher Values Indicate: Increased treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Husnu Efendi, Prof., Study Chair — Kocaeli University; Mehmet Fatih Yetkin Assoc. Prof. MD, Assoc. Prof., Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 3 years after the publication of results

REFERENCES:
- [Background] Comi G, Freedman MS, Meca-Lallana JE, Vermersch P, Kim BJ, Parajeles A, Edwards KR, Gold R, Korideck H, Chavin J, Poole EM, Coyle PK. Prior treatment status: impact on the efficacy and safety of teriflunomide in multiple sclerosis. BMC Neurol. 2020 Oct 6;20(1):364. doi: 10.1186/s12883-020-01937-4. PMID 33023488
- [Background] Berkovich R, Negroski D, Wynn D, Sellers D, Bzdek KG, Lublin AL, Rawlings AM, Quach C, Wells DP, Dumlao M, Bora A, Ranno AE, Luo KL, Chavin J, Hua LH, Becker D. Effectiveness and safety of switching to teriflunomide in older patients with relapsing multiple sclerosis: A real-world retrospective multicenter analysis. Mult Scler Relat Disord. 2023 Feb;70:104472. doi: 10.1016/j.msard.2022.104472. Epub 2022 Dec 18. PMID 36566698
- [Background] Bencsik K, Dobos E, Jobbagy Z, Birkas AJ, Kovacs K, Satori M, Lencses G, Bartok G, Losonczi E, Vecsei L, On Behalf Of The Teri-Real Investigators. Real-World Evidence for Favourable Quality-of-Life Outcomes in Hungarian Patients with Relapsing-Remitting Multiple Sclerosis Treated for Two Years with Oral Teriflunomide: Results of the Teri-REAL Study. Pharmaceuticals (Basel). 2022 May 13;15(5):598. doi: 10.3390/ph15050598. PMID 35631424
- [Background] Elkhooly M, Bao F, Bernitsas E. Impact of Disease Modifying Therapy on MS-Related Fatigue: A Narrative Review. Brain Sci. 2023 Dec 20;14(1):4. doi: 10.3390/brainsci14010004. PMID 38275509
- [Background] Meca-Lallana JE, Prieto Gonzalez JM, Caminero Rodriguez AB, Olascoaga Urtaza J, Alonso AM, Duran Ferreras E, Espinosa R, Dotor J, Romera M, Ares Luque A, Perez Ruiz D, Calles C, Hernandez MA, Hervas Garcia M, Mendoza Rodriguez A, Berdei Montero Y, Tellez N, Herrera Varo N, Sotoca J, Presas-Rodriguez S, Querol Gutierrez LA, Hervas Pujol M, Batlle Nadal J, Martin Ozaeta G, Gubieras Lillo L, Martinez Yelamos S, Ramio-Torrenta L, Mallada Frechin J, Belenguer Benavides A, Gascon-Gimenez F, Casanova B, Landete Pascual L, Berenguer L, Navarro L, Gomez Gutierrez M, Duran C, Rodriguez Regal A, Alvarez E, Garcia-Estevez DA, Lopez Real AM, Llaneza Gonzalez MA, Marzo Sola ME, Sanchez-Menoyo JL, Oterino A, Villaverde Gonzalez R, Castillo-Trivino T, Alvarez de Arcaya A, Llarena C. Effectiveness and Safety of Teriflunomide in Relapsing-Remitting Multiple Sclerosis and Improvements in Quality of Life: Results from the Real-World TERICARE Study. Neurol Ther. 2023 Dec;12(6):2177-2193. doi: 10.1007/s40120-023-00557-7. Epub 2023 Oct 20. PMID 37861931
- [Background] Strosova D, Tuzil J, Turkova BV, Pilnackova BF, de Souza LL, Dolezalova H, Raskova M, Dufek M, Dolezal T. Relationship between Patient Preferences, Attitudes to Treatment, Adherence, and Quality of Life in New Users of Teriflunomide. Pharmaceuticals (Basel). 2022 Oct 11;15(10):1248. doi: 10.3390/ph15101248. PMID 36297360
- [Background] Miller AE. An updated review of teriflunomide's use in multiple sclerosis. Neurodegener Dis Manag. 2021 Oct;11(5):387-409. doi: 10.2217/nmt-2021-0014. Epub 2021 Sep 16. PMID 34486382
- [Background] Coyle PK, Khatri B, Edwards KR, Meca-Lallana JE, Cavalier S, Rufi P, Benamor M, Thangavelu K, Robinson M, Gold R; Teri-PRO Trial Group. Patient-reported outcomes in patients with relapsing forms of MS switching to teriflunomide from other disease-modifying therapies: Results from the global Phase 4 Teri-PRO study in routine clinical practice. Mult Scler Relat Disord. 2018 Nov;26:211-218. doi: 10.1016/j.msard.2018.09.017. Epub 2018 Sep 15. PMID 30273841
- [Background] Hestvik ALK, Frederiksen JL, Nielsen HH, Torkildsen O, Eek C, Huang-Link Y, Haghighi S, Tsai JA, Kant M. Real-world study of relapsing-remitting multiple sclerosis patients treated with Teriflunomide in Nordic countries: Quality-Of-Life, efficacy, safety and adherence outcomes. Mult Scler Relat Disord. 2022 Jul;63:103892. doi: 10.1016/j.msard.2022.103892. Epub 2022 May 16. PMID 35696880
- [Background] de Seze J, Devy R, Planque E, Delabrousse-Mayoux JP, Vandhuick O, Kabir M, Gherib A. Fatigue in teriflunomide-treated patients with relapsing remitting multiple sclerosis in the real-world Teri-FAST study. Mult Scler Relat Disord. 2021 Jan;47:102659. doi: 10.1016/j.msard.2020.102659. Epub 2020 Nov 28. PMID 33291032
- [Background] Garnock-Jones KP. Teriflunomide: a review of its use in relapsing multiple sclerosis. CNS Drugs. 2013 Dec;27(12):1103-23. doi: 10.1007/s40263-013-0118-2. PMID 24198223